CLINICAL TRIAL: NCT04495855
Title: VISANNE OS/Treatment of Endometriosis With Dienogest in the Real World Clinical Practice
Brief Title: A Study to Learn More About Using Dienogest to Treat Endometriosis in Chinese Participants
Acronym: VISANNE OS
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 21088
Record Dates: First submitted 2020-07-14; First posted 2020-08-03 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Endometriosis
MeSH Terms: conditions — Endometriosis | interventions — dienogest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Visanne treatment: Patients from post-menarche to menopause with clinically or surgically diagnosed endometriosis, who have been prescribed Visanne
  Interventions: Drug: Dienogest (Visanne,BAY86_5258)

INTERVENTIONS:
Drug: Dienogest (Visanne,BAY86_5258) — 2 mg (once a day), oral, tablet.

SUMMARY:
Endometriosis is a condition that affects women, usually during their reproductive years. In women with endometriosis, the tissue that lines the uterus starts to grow outside of the uterus. This can cause pain during their periods or during sex, and constant pain in the pelvis. Endometriosis can decrease a woman's quality of life and requires long-term treatment to control the symptoms.

For some women with endometriosis, symptoms can return after they stop treatment. Or, they may not be able to tolerate the current long-term treatment options.

In this study, researchers will find out more about the safety of long-term treatment with dienogest in a large number of Chinese participants. This study will enroll patients from post-menarche to menopause with clinically or surgically diagnosed endometriosis. All of the participants will take dienogest based on their doctor's instructions. They will then visit their doctor's office 3 times over 6 months. During these visits, their doctors will ask them if they have any health problems and about their quality of life. Their doctors will also do tests to measure the pain caused by their endometriosis and any other symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent.
* Post-menarcheal age through menopause.
* Have clinically or surgically diagnosed endometriosis according to routine clinical practice.
* Decision for the treatment with Visanne was made as per physician's routine treatment practice.

Exclusion Criteria:

* Patients participating in an investigational program with interventions outside of routine clinical practice.
* Any contraindication according to Visanne Chinese label

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Chinese patients from post-menarche to menopause diagnosed with endometriosis, either surgically or clinically, and prescribed with Visanne by a physician according to China's health authority approved label.
Sampling Method: Non-Probability Sample
Enrollment: 968 (Actual)
Dates: Start 2020-10-28 (Actual); Primary Completion 2022-12-23 (Actual); Study Completion 2022-12-23 (Actual)

PRIMARY OUTCOMES:
The absolute number of AEs reported with Visanne treatment | From baseline up to 6 months
  AE: Adverse Event
The absolute number of ADRs reported with Visanne treatment | From baseline up to 6 months
  ADR: Adverse drug reaction
The proportion of AEs reported with Visanne treatment | From baseline up to 6 months
  Proportion of each AE will be calculated as number of patients with at least one event divided by the total number of patients.
The proportion of ADRs reported with Visanne treatment | From baseline up to 6 months
  Proportion of each ADR will be calculated as number of patients with at least one event divided by the total number of patients.

SECONDARY OUTCOMES:
Changes in Numeric Rating Scale (NRS) score of Endometriosis Associated Pelvic Pain (EAPP) of Visanne treatment | From baseline up to 1,3,6 months
  NRS: 0-10 integers."absence of pain" corresponds to the value of "0" and unbearable pain corresponding to the value of "10".
Endometriosis Health Profile-5 (EHP-5) score changes with Visanne treatment | At baseline and 6 months.
  EHP-5 contains 11 questions (items): five items including pain, control and powerlessness, emotional well-being, lack of social support, self image from the core questionnaire and six items from the modular questionnaire that may not be applicable to every woman with endometriosis including work, intercourse, and worries about infertility, treatment, and relationship with children and medical professionals. Each item is rated on a four-point scale (never = 0, rarely = 1, sometimes = 2, often = 3, always = 4 and not relevant if not applicable).
Patient and physician's satisfaction score on Visanne® treatment | At 3 and 6 months
  Satisfaction will be assessed in 5 scales (very satisfied, somewhat satisfied, neither satisfied or dissatisfied, somewhat dissatisfied, very dissatisfied)
Changes in Clinical Global Impression (CGI) scale scores of overall symptom development | At 3 and 6 months
  CGI scale: very much improved, much improved, minimally improved, no change, minimally worse, much worse, very much worse
Changes in Patient Global Impression (PGI-C) scale scores of overall symptom development | At 3 and 6 months
  PGI-C scale: very much improved, much improved, minimally improved, no change, minimally worse, much worse, very much worse
Reasons for discontinuation of using Visanne | From baseline up to 6 months
  Discontinuation reasons identification:
  * AEs (Exclude expected menstruation and treatment ineffective)
  * Dissatisfaction with bleeding profile
  * Absence of symptoms
  * Treatment ineffective
  * Physicians decision
  * Switching to another treatment (another medicine or surgery)
  * Wish to conceive
  * Others
The proportion of participant with amenorrhea, infrequent bleeding, frequent bleeding irregular bleeding, prolonged bleeding upon treatment with Visanne | At baseline, 1, 3, and 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Many locations, Multiple Locations, China

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.